CLINICAL TRIAL: NCT01244165
Title: Clinical Investigation of Fetal Bovine Dermis Material (Cytrix) for Use in the Treatment of Pelvic Floor Prolapse
Brief Title: Study of Cytrix Use in Pelvic Floor Prolapse Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Janice Connor / Director, Clinical Affairs, Boston Scientific
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WH-2004-01
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Vaginal Vault Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cytrix (Other): Observational Study
  Interventions: Device: Cytrix
- Control Group (Other): Patients with similar indications who were treated at the same centers using other products
  Interventions: Other: Other treatments for pelvic organ prolapse

INTERVENTIONS:
Device: Cytrix
  Arms: Cytrix
Other: Other treatments for pelvic organ prolapse — Treatments for pelvic organ prolapse using other products (standard of care for treatment of pelvic organ prolapse)
  Arms: Control Group

SUMMARY:
To evaluate safety and effectiveness of using the fetal bovine dermis (Cytrix) in the treatment of pelvic organ prolapse.

ELIGIBILITY:
Inclusion Criteria:

* Female >30 years of age
* Willing and able to comply w/ the study procedures and provide written informed consent to participate in the study.
* Diagnosed with pelvic organ prolapse with or without pelvis floor dysfunction
* Patient is willing to complete PFDI-SF20 and PISQ-12 questionnaires at 6 and 12 months post-operatively
* Patient is willing to answer phone questionnaires at 2 weeks, 6 weeks, and 3 months
* Patients with a history of pelvic surgery (cystocele/anterior repair, hysterectomy, vault suspension, etc) prior to this procedure are allowed to participate in the study except if the patient had a dermal graft implanted.

Exclusion Criteria:

* Patients who, in the clinical judgment of the investigator, are not suitable for this study
* Patients who are, in the Investigators opinion, mentally or legally incapacitated preventing informed consent or unable to read or understand written material.
* Patients who have participated in an investigational study within 30 days of study entry that may impact analysis of this device or have previously participated in the current trial
* Patient whose pelvic organ prolapse is Stage I
* Patient with Diabetes Mellitus type I or II
* Patient with morbid obesity (weight parameters determined by physician)
* Patient with undiagnosed pelvic mass outside of the uterus (not expected to be functional in nature)
* Patient with unexplained abnormal menstrual bleeding
* Patient with any acute or chronic infection (kidney, bladder, lung, etc)
* Patient with coagulopathy
* Patient participating in other investigational device or drug study
* Patients must not be pregnant
* Patients with life expectancy less than 2 years
* Patients with known or suspected hypersensitivity to collagen or bovine products
* Patients with preexisting local or systemic infection
* Patients with a history of soft tissue pathology where the implant is to be placed
* Patients with any pathology that would limit the blood supply and compromise healing
* Patient diagnosed with autoimmune connective tissue disease

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2002-01; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Number of patients reporting intra-operative complications | at procedure
number of treated patients reporting post-operative adverse events | 6 Months
Patient healing time | 6 Months
  length of hospital stay and pain medication
Incidence of complication in Cytrix treated patients compared to patients in the historical control group | 6 months
  Incidence of complication in Cytrix treated patients compared to patients in the historical control group
Patient satisfaction after Pelvic Organ Prolapse surgery using Cytrix | 3 months
  Phone-Patient Questionnaire
Patient satisfaction after Pelvic Organ Prolapse surgery using Cytrix | 6 months
  Pelvic Floor Distress Inventory (PFDI-SF20) Patient questionnaire, and Pelvic Organ Prolapse Sexual Questionnaire (PISQ-12) Questionnaire
Patient satisfaction after Pelvic Organ Prolapse surgery using Cytrix | 12 months
Comparison of phone patient questionnaire results between Cytrix Group and Control Group | 6 months
  Comparison of phone patient questionnaire results in Cytrix treated patients compared to patients in the retrospective historical control group where available.
Patient satisfaction after Pelvic Organ Prolapse surgery using Cytrix | 2 wks
  Phone-Patient Questionnaire
Patient satisfaction after Pelvic Organ Prolapse surgery using Cytrix | 6 wks
  Phone-Patient Questionnaire
Comparison of Pelvic Floor Distress Inventory (PFDI-SF20) questionnaire results between Cytrix Group and Control Group | 6 months
  Comparison of Pelvic Floor Distress Inventory (PFDI-SF20) questionnaire results in Cytrix treated patients compared to patients in the retrospective historical control group where available.

SECONDARY OUTCOMES:
Physician satisfaction in the treatment of patients with pelvic floor prolapse using Cytrix | 6 months
  Physician satisfaction in the treatment of patients with pelvic floor prolapse using Cytrix versus any other product currently being the standard method of care;
  1. handling characteristics
  2. conformity to the surgical site
  3. ease of suture
  4. procedure length of time

CONTACTS AND LOCATIONS:
Overall Officials: Oscar A Aguirre, MD, Principal Investigator — Milestone Medical Research

REFERENCES:
- [Derived] Goldstein HB, Maccarone J, Naughton MJ, Aguirre OA, Patel RC. A multicenter prospective trial evaluating fetal bovine dermal graft (Xenform(R) Matrix) for pelvic reconstructive surgery. BMC Urol. 2010 Dec 13;10:21. doi: 10.1186/1471-2490-10-21. PMID 21144043